CLINICAL TRIAL: NCT02922465
Title: Drug-Drug Interaction Study to Assess the Effects of Multi Dose Clopidogrel on the Pharmacokinetics of Single-Dose K-877 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: K-877-109
Record Dates: First submitted 2016-09-15; First posted 2016-10-04 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Healthy
MeSH Terms: interventions — K-877 compound; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- K-877 & Clopidogrel (Experimental): K-877 & Clopidogrel orally
  Interventions: Drug: K-877; Drug: Clopidogrel

INTERVENTIONS:
Drug: K-877
Drug: Clopidogrel

SUMMARY:
The primary objective of this study is to assess the effects of clopidogrel on the PK of K-877 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject provides written informed consent before any study-specific evaluation is performed;
* Subject is a healthy adult male or female volunteer between the ages of 18 and 45 years, inclusive at screening;
* Subject has a BMI of 18 to 30 kg/m², inclusive;
* Subject has hematology, serum chemistry, and urinalysis test results within the reference ranges, or results that do not show clinically significant abnormalities, as judged by the Investigator at screening and check-in;

Exclusion Criteria:

* Subject is a woman who is pregnant or breastfeeding;
* Subject has clinically significant abnormalities in the screening or check-in assessments;
* Subject has current or history of clinically significant coagulation, bleeding, or platelet disorders;
* Subject or a family member of the subject has a history of coagulation or bleeding disorders or reasonable suspicion of vascular malformations, including aneurysms;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Plasma exposure of K-877 by measuring Cmax when administered alone or with Clopidogrel | Up to 72 hours after dosing
Plasma exposure of K-877 by measuring AUC when administered alone or with Clopidogrel | Up to 72 hours after dosing

SECONDARY OUTCOMES:
Evaluation of 20 participants with treatment emergent adverse events as assessed by the principle investigator | Through study completion up to 17 days.
  Subjects will be questioned in a general way by the investigator without specific symptoms suggested.

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati, Ohio, United States